CLINICAL TRIAL: NCT00665093
Title: A Prospective, Multicentre, Open Label, Non-controlled, Observational, 24-week Study in Patients Using NovoMix® 30 (Biphasic Insulin Aspart 30) or Levemir® (Insulin Detemir) for Treatment of Type 1 or Type 2 Diabetes Mellitus in Macedonia
Brief Title: Observational Study of Patients Using NovoMix® 30 or Levemir® for Treatment of Type 1 or Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-1894
Record Dates: First submitted 2008-04-22; First posted 2008-04-23 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A
  Interventions: Drug: biphasic insulin aspart 30
- B
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Start dose and frequency prescribed by the physician as a result of a normal clinical evaluation
  Other Names: NovoMix® 30; BIASP
  Groups: A
Drug: insulin detemir — Start dose and frequency prescribed by the physician as a result of a normal clinical evaluation
  Groups: B

SUMMARY:
This trial is conducted in Europe. The aim of this observational study is to evaluate the glycaemic control in patients with type 1 or 2 diabetes using NovoMix® 30 or Levemir® under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Levemir® above 6 yrs
* NovoMix® 30 above 18 yrs
* Patients with Type 1 or Type 2 diabetes, including newly diagnosed

Exclusion Criteria:

* Current treatment with NovoMix® 30 or Levemir®

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 1 and Type 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 1569 (Actual)
Dates: Start 2007-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
HbA1c | at 24 weeks

SECONDARY OUTCOMES:
FPG, PG profile, weight, % of subjects on target | at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Skopje, North Macedonia

REFERENCES:
- [Result] Milenkovic T. Significant Improvements in Glycemic Control with BIAsp 30 in Clinical Reality: Experience from clinical practice in Macedonia. ADA American Diabetes Association 2009; Country: USA City: New Orleans
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com